CLINICAL TRIAL: NCT05687903
Title: A Randomized, Double-blind, Placebo-Controlled Study to Evaluate the Efficacy, Safety, and Tolerability of TAK-861 for the Treatment of Narcolepsy With Cataplexy (Narcolepsy Type 1)
Brief Title: A Study of TAK-861 in Participants With Narcolepsy Type 1
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: TAK-861-2001; 2022-001654-38 (EudraCT Number); U1111-1277-4261 (Other: WHO); jRCT2031220644 (Registry Identifier: jRCT)
Record Dates: First submitted 2023-01-09; First posted 2023-01-18 (Actual); Results first posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2024-12

CONDITIONS: Narcolepsy Type 1
Keywords: Drug Therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Placebo (Placebo Comparator): Participants received placebo tablets matching TAK-861, orally, twice daily (BID), from Days 1 to 56.
  Interventions: Drug: Placebo
- TAK-861 0.5 mg BID (Experimental): Participants received TAK-861 0.5 milligrams (mg), orally, BID, from Days 1 to 56.
  Interventions: Drug: TAK-861
- TAK-861 2 mg BID (Experimental): Participants received TAK-861 2 mg, orally, BID, from Days 1 to 56.
  Interventions: Drug: TAK-861
- TAK-861 2 mg and 5 mg (Experimental): Participants received TAK-861 2 mg followed by 5 mg dose, orally, BID, from Days 1 to 56.
  Interventions: Drug: TAK-861
- TAK-861 7 mg QD (Experimental): Participants received TAK-861 7 mg, orally, once daily (QD), from Day 1 to 56. Placebo was given as the second dose.
  Interventions: Drug: TAK-861; Drug: Placebo

INTERVENTIONS:
Drug: TAK-861 — TAK-861 oral tablets
  Arms: TAK-861 0.5 mg BID; TAK-861 2 mg BID; TAK-861 2 mg and 5 mg; TAK-861 7 mg QD
Drug: Placebo — Placebo oral tablets matching TAK-861
  Arms: Placebo; TAK-861 7 mg QD

SUMMARY:
The main aim of this study is to see how TAK-861 works on symptoms of narcolepsy, including excessive daytime sleepiness and cataplexy. Approximately 100 participants will take part in the study across North America, Europe and Asia Pacific.

The treatment (TAK-861 or placebo) will be administered for 8 or 12 weeks. After this treatment period the participant will have the option to participate in a separate, long- term extension study during which all participants will be treated with TAK-861.

DETAILED DESCRIPTION:
The drug being tested in this study is called TAK-861. This study will look at the effect of TAK-861 on improvement in narcolepsy symptoms, including excessive daytime sleepiness (EDS) and number of cataplexy episodes.

The study will enroll approximately 100 patients. Participants will be randomly assigned (by chance, like flipping a coin) to one of the five treatment groups which will remain undisclosed to the participant and study doctor during the study (unless there is an urgent medical need):

* TAK-861 Dose 1
* TAK-861 Dose 2
* TAK-861 Dose 3
* TAK-861 Dose 4
* Placebo (dummy inactive pill) - this is a tablet that looks like the study drug but has no active ingredient

This multi-center trial will be conducted worldwide. The overall time to participate in this study is up to 23 weeks. Participants will make multiple visits to the clinic during the treatment period and then will either enroll in a long-term extension study in which all participants will receive TAK-861 or have 2 final visits 7 and 28 days after last dose of study drug for follow-up assessments.

ELIGIBILITY:
Inclusion Criteria:

1. The participant is aged 18 to 70 years, inclusive, at the time of signing the informed consent form (ICF).

   Note: In Japan, participants aged 16 to 70 years, inclusive, may be included.
2. The participant has body mass index (BMI) within the range 18 to 40 kilogram per square meter [kg/m^2] (inclusive).
3. The participant has an International Classification of Sleep Disorders, 3rd Edition (ICSD-3) diagnosis of narcolepsy type 1 (NT1) by polysomnography (PSG)/Multiple Sleep Latency Test (MSLT), performed within the past 10 years.
4. The participant is positive for the human leukocyte antigen (HLA) genotype HLA-DQB1*06:02 or results from cerebrospinal fluid (CSF) testing indicate the participant's CSF orexin (OX)/hypocretin-1 concentration is <110 picograms per milliliter ([pg/mL] (or less than one-third of the mean values obtained in normal participants within the same standardized assay).

Exclusion Criteria:

1. The participant has a current medical disorder, other than narcolepsy with cataplexy, associated with EDS.
2. The participant has medically significant hepatic or thyroid disease.
3. The participant has a history of cancer in the past 5 years (does not apply to participants with carcinoma in situ that has been resolved without further treatment or basal cell cancer).
4. The participant has clinically significant coronary artery disease, a history of myocardial infarction, clinically significant angina, clinically significant cardiac rhythm abnormality, or heart failure.
5. The participant has a clinically significant history of head injury or head trauma.
6. The participant has history of epilepsy, seizure, or convulsion, or has a family history of inherited disorders associated with seizure (except for a single febrile seizure in childhood).
7. The participant has one or more of the following psychiatric disorders:

   1. Any current unstable psychiatric disorder.
   2. Current or history of manic or hypomanic episode, schizophrenia or any other psychotic disorder, including schizoaffective disorder, major depression with psychotic features, bipolar depression with psychotic features, obsessive compulsive disorder, intellectual disability, organic mental disorders, or mental disorders due to a general medical condition as defined in the Diagnostic and Statistical Manual of Mental Disorders, 5th Edition (DSM-5).
   3. Current diagnosis or history of substance use disorder as defined in the DSM-5.
   4. Current active major depressive episode (MDE) or who have had an active MDE in the past 6 months.
8. The participant has a history of cerebral ischemia, transient ischemic attack (<5 years ago), intracranial aneurysm, or arteriovenous malformation.
9. The participant has a positive test result for hepatitis B surface antigen, hepatitis C virus antibody, or human immunodeficiency virus (HIV) antibody/antigen.
10. The participant's renal creatinine clearance (Cockcroft-Gault Equation) is ≤50 mL/minute.
11. The participant has alanine aminotransferase (ALT) or aspartate aminotransferase (AST) values >1.5 times the upper limit of normal (ULN).
12. The participant is considered by the investigator to be at imminent risk of suicide or injury to self, others, or property, or the participant has attempted suicide within the past year.

Ages: 16 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 112 (Actual)
Dates: Start 2023-01-09 (Actual); Primary Completion 2023-12-14 (Actual); Study Completion 2023-12-14 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (57):
- United States (21):
  - Sleep Disorders Center of Alabama, Birmingham, Alabama
  - Stanford Center for Sleep Sciences and Medicine, Redwood City, California
  - SDS Clinical Trials, Inc., Santa Ana, California
  - Delta Waves LLC - Hunt - PPDS, Sleep Disorder and Research Center, Colorado Springs, Colorado
  - Florida Pediatric Research Institute, Orlando, Florida
  - Neurotrials Research, Atlanta, Georgia
  - Georgia Neuro Center, Gainesville, Georgia
  - University of Kansas Medical Center Research Institute, Inc., Kansas City, Kansas
  - Neurocare Inc, Newton, Massachusetts
  - Henry Ford Medical Center - Columbus, Novi, Michigan
  - St. Lukes Sleep Medicine and Research Center, Chesterfield, Missouri
  - Research Carolina Elite, Denver, North Carolina
  - ARSM Research, LLC, Huntersville, North Carolina
  - Intrepid Research, Cincinnati, Ohio
  - The Cleveland Clinic Foundation, Cleveland, Ohio
  - Ohio Sleep Medicine Institute, Dublin, Ohio
  - Medical University of South Carolina - PPDS, Charleston, South Carolina
  - Bogan Sleep Consultants, LLC, Columbia, South Carolina
  - Comprehensive Sleep Medicine Associates - Sugar Land, Houston, Texas
  - Sleep Therapy and Research Center, San Antonio, Texas
  - Children's Specialty Group, Norfolk, Virginia
- Woolcock Institute of Medical Research, Sleep and Circadian Research Group, Glebe, New South Wales, Australia
- Terveystalo Helsinki Sleep Clinic, Helsinki, Uusimaa, Finland
- France (4):
  - Hopital Pierre-Paul Riquet, Toulouse, Haute-Garonne
  - CHU Gui De Chauliac, Montpellier, Herault
  - CHU de Grenoble, La Tronche, Isere
  - Hopital de la Pitie Salpetriere, Paris
- Germany (4):
  - Universitaet Regensburg am Bezirksklinikum, Regensburg, Bavaria
  - Somni Bene Institut fur Medizinische Forschung und Schlafmedizin Schwerin GmbH, Schwerin, Mecklenburg-Vorpommern
  - Charite - Universitatsmedizin Berlin, Berlin
  - Klinische Forschung Hamburg, Hamburg
- Italy (3):
  - IRCCS Istituto delle Scienze Neurologiche di Bologna, Dipartimento di Scienze Biomediche e Neuromotorie, Bellaria, Bologna
  - Fondazione PTV Policlinico Tor Vergata, Centro del Sonno e del Trattamento Neurologico delle Fragilta, Rome, Lazio
  - Istituto Neurologico Mediterraneo Neuromed, Centro Per La Diagnosi E la Cura Del Sonno, Pozzilli, Molise
- Japan (9):
  - Akita University Hospital, Akita, Akita
  - Kurume University Hospital, Kurume-Shi, Hukuoka
  - Howakai Kuwamizu Hospital, Chuo-Ku, Kumamoto, Kumamoto
  - Gokeikai Osaka Kaisei Hospital, Yodogawa-Ku, Osaka, Osaka
  - Koishikawa Tokyo Hospital, Bunkyo-Ku, Tokyo
  - National Center of Neurology and Psychiatry, Kodaira-Shi, Tokyo
  - Yoyogi Sleep Disorder Center, Shibuya-Ku, Tokyo
  - Aichi Medical University Hospital, Nagakute
  - RESM respiratory and sleep medical-care clinic, Yokoharna Building, 4Floor, Yokohama
- Netherlands (2):
  - Kempenhaeghe - PPDS, Heeze, North Brabant
  - Slaap-Waakcentrum SEIN Heemstede, Heemstede, North Holland
- University of Oslo, Oslo, Norway
- Spain (7):
  - Hospital Universitario Araba Santiago, Unidad Funcional de Sueno, Vitoria-Gasteiz, Alava
  - Hospital General de Castello, Sleep Unit, Castellon, Castellon
  - Hospital de La Ribera, Unidad de Sueno, Alzira, Valencia
  - Hospital Universitario Vall d'Hebron - PPDS, Barcelona
  - Hospital Clinic de Barcelona, Neurology Service, scale 8-4th floor, Barcelona
  - Instituto de Investigaciones del Sueno, Madrid
  - Hospital Vithas Madrid Arturo Soria, Madrid
- Sahlgrenska Universitetssjukhuset, Gothenburg, Västra Götaland County, Sweden
- Switzerland (3):
  - Klinik Barmelweid AG, Barmelweid, Aargau (de)
  - Neurocenter of Southern Switzerland, Lugano, Ticino (it)
  - Universitaetsspital Bern, Department of Neurology, Bern

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/. For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- [Derived] Lammers GJ, Plazzi G, Mignot E, Pizza F, Dauvilliers Y, Barateau L, Maruff P, Scammell TE, Latzman RD, Naylor M, Olsson T, Stukalin E, Tanaka S, Volfson D, Khachadourian V, Harel BT. Effects of Oveporexton, an Orexin Receptor 2-Selective Agonist, on Cognition in Narcolepsy Type 1: A Secondary Analysis of a Randomized Clinical Trial. JAMA Neurol. 2025 Dec 8:e254825. doi: 10.1001/jamaneurol.2025.4825. Online ahead of print. PMID 41359331
- [Derived] Dauvilliers Y, Plazzi G, Mignot E, Lammers GJ, Del Rio Villegas R, Khatami R, Taniguchi M, Abraham A, Hang Y, Kadali H, Lamberton M, Sheikh S, Stukalin E, Neuwirth R, Swick TJ, Tanaka S, von Hehn C, von Rosenstiel P, Wang H, Cai A, Naylor M, Olsson T. Oveporexton, an Oral Orexin Receptor 2-Selective Agonist, in Narcolepsy Type 1. N Engl J Med. 2025 May 15;392(19):1905-1916. doi: 10.1056/NEJMoa2405847. PMID 40367374
- See also: To obtain more information on the study, click here/on this link — https://clinicaltrials.takeda.com/study-detail/4c5a5e765b46449e?idFilter=%5B%22TAK-861-2001%22%5D

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study at 33 investigative sites globally from 09 January 2023 to 14 December 2023.
Pre-assignment Details: Participants with a diagnosis of narcolepsy type 1 (NT1) were enrolled in the study to receive either TAK-861 or placebo.
Groups:
- TAK-861 2 mg and 5 mg: Participants received TAK-861 2 mg followed by the 5 mg dose, orally, from Days 1 to 56.
- TAK-861 7 mg QD: Participants received TAK-861 7 mg, orally, once daily (QD), from Days 1 to 56. Placebo was given as the second dose.
Period: Overall Study
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD
Started | 22 | 23 | 21 | 23 | 23
Completed | 21 | 22 | 21 | 22 | 23
Not Completed | 1 | 1 | 0 | 1 | 0
Not completed — Protocol Deviation | 1 | 1 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Groups:
- Placebo: Participants received placebo tablets matching TAK-861, orally, BID, from Days 1 to 56.
- TAK-861 0.5 mg BID: Participants received TAK-861 0.5 mg, orally, BID, from Days 1 to 56.
- TAK-861 7 mg QD: Participants received TAK-861 7 mg, orally, QD, from Days 1 to 56. Placebo was given as the second dose.
- Total: Total of all reporting groups
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD | Total
Number analyzed (Participants) | 22 | 23 | 21 | 23 | 23 | 112
Age, Continuous [Mean (Standard Deviation); unit: years] | 37.5 (11.86) | 32.7 (11.06) | 31.7 (11.31) | 34.7 (11.48) | 33.3 (11.94) | 34 (11.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 11 | 9 | 14 | 10 | 58
  Male | 8 | 12 | 12 | 9 | 13 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 2 | 1 | 0 | 2 | 8
  Not Hispanic or Latino | 19 | 21 | 20 | 23 | 20 | 103
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 1 | 2 | 0 | 3 | 2 | 8
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 2 | 1 | 2 | 0 | 1 | 6
  White | 19 | 19 | 19 | 19 | 20 | 96
  More than one race | 0 | 1 | 0 | 1 | 0 | 2
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Average Sleep Latency From the Maintenance of Wakefulness Test (MWT) [Mean (Standard Deviation); unit: minutes] — The MWT is a validated, objective measure that evaluates a participant's ability to remain awake under soporific conditions for a defined period. During each MWT session (1 session = 40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on electroencephalography (EEG). If no sleep was observed according to these rules, then the latency was defined as 40 minutes. Population: Number analyzed is the number of participants with data available for analyses at Baseline.
  minutes
    number analyzed (Participants) | 22 | 23 | 21 | 22 | 23 | 111
    (all) | 6.1 (8.82) | 5.6 (7.89) | 3.9 (5.98) | 4.2 (3.63) | 3.6 (4.87) | 4.7 (6.48)

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in the Average Sleep Latency as Determined From the MWT at Week 8
Description: The MWT is a validated, objective measure that evaluates a participant's ability to remain awake under soporific conditions for a defined period. During each MWT session (1 session = 40 minutes), participants were instructed to sit quietly and remain awake for as long as possible. Sleep latency in each session was recorded on EEG. If no sleep was observed according to these rules, then the latency was defined as 40 minutes. The linear mixed effects model for repeated measures (MMRM) was used for analysis.
Time Frame: Baseline, Week 8
Population: Full Analysis Set included all participants who were randomized and received at least one dose of study drug and had at least one post-dose efficacy measurement. Overall number of participants analyzed is the number of participants with data available for analyses.
Measure: Least Squares Mean (Standard Error); unit: minutes
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD
Number analyzed (Participants) | 21 | 19 | 21 | 20 | 23
minutes | -1.16 (2.061) | 12.49 (2.128) | 23.50 (2.042) | 25.42 (2.071) | 14.96 (1.953)
Statistical Analysis 1: Comparison: Placebo vs TAK-861 0.5 mg BID; Test type: Superiority; p = 0.001, MMRM — The analysis used a linear MMRM with fixed effects for Baseline, age, prior use of narcolepsy medications, treatment, visit, and treatment-by-visit interaction as covariates. Reported p-value is adjusted for multiplicity; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = 13.65, 95% CI 2-sided [7.74 to 19.57], Standard Error of Mean 2.983 — LS in LS Mean Difference denotes least squares
Statistical Analysis 2: Comparison: Placebo vs TAK-861 2 mg BID; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = 24.67, 95% CI 2-sided [18.87 to 30.46], Standard Error of Mean 2.921
Statistical Analysis 3: Comparison: Placebo vs TAK-861 2 mg and 5 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = 26.58, 95% CI 2-sided [20.81 to 32.35], Standard Error of Mean 2.91
Statistical Analysis 4: Comparison: Placebo vs TAK-861 7 mg QD; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = 16.13, 95% CI 2-sided [10.49 to 21.76], Standard Error of Mean 2.842

2. Secondary Outcome: Change From Baseline in Epworth Sleepiness Scale (ESS) Total Score at Week 8
Description: The ESS is a subjective, self-administered, validated scale (scored 0 to 3) to respond to each of the 8 questions of daily life that asks participants how likely they are to fall asleep in those situations. The scores are summed to give an overall score of 0 to 24. Higher scores indicate stronger subjective daytime sleepiness, and scores below 10 are considered to be within the normal range. The MMRM was used for analysis.
Time Frame: Baseline, Week 8
Population: as for outcome 1
Measure: Least Squares Mean (Standard Error); unit: score on a scale
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD
Number analyzed (Participants) | 21 | 21 | 21 | 22 | 23
score on a scale | -2.50 (1.109) | -8.92 (1.085) | -13.79 (1.115) | -12.81 (1.073) | -11.29 (1.064)
Statistical Analysis 1: Comparison: Placebo vs TAK-861 0.5 mg BID; Test type: Superiority; p = 0.004, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = -6.42, 95% CI 2-sided [-9.53 to -3.32], Standard Error of Mean 1.564
Statistical Analysis 2: Comparison: Placebo vs TAK-861 2 mg BID; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = -11.3, 95% CI 2-sided [-14.44 to -8.16], Standard Error of Mean 1.581
Statistical Analysis 3: Comparison: Placebo vs TAK-861 2 mg and 5 mg; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = -10.31, 95% CI 2-sided [-13.35 to -7.27], Standard Error of Mean 1.53
Statistical Analysis 4: Comparison: Placebo vs TAK-861 7 mg QD; Test type: Superiority; p < 0.001, MMRM — [p-value comment as in outcome 1, analysis 1]; An unstructured variance-covariance structure was used; Estimate of LS Mean Difference = -8.79, 95% CI 2-sided [-11.84 to -5.75], Standard Error of Mean 1.535

3. Secondary Outcome: Weekly Cataplexy Rate (WCR) at Week 8
Description: Participants completed a daily patient-reported sleep diary to record self-reported narcolepsy symptoms. Participants recorded episodes of cataplexy attacks in the diary. The total number of events averaged for a week were reported. WCR = (total number of cataplexy attacks over a number of non-missing diary days for a given duration/number of non-missing diary days in that duration)*7. The generalized estimating equations (GEE) model was used for analysis.
Time Frame: Week 8
Population: as for outcome 1
Measure: Least Squares Mean (95% Confidence Interval); unit: cataplexy attacks per week
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD
Number analyzed (Participants) | 20 | 21 | 21 | 22 | 23
cataplexy attacks per week | 8.76 [5.68 to 13.51] | 4.24 [2.60 to 6.92] | 3.14 [1.65 to 5.98] | 2.48 [1.30 to 4.73] | 5.89 [3.64 to 9.53]
Statistical Analysis 1: Comparison: Placebo vs TAK-861 0.5 mg BID; The GEE model was used for analysis with fixed effects for visit, treatment, treatment-by-visit interaction, Baseline WCR, age, and prior use of narcolepsy medications; Test type: Superiority; p = 0.250, GEE — GEE model featuring a negative binomial distribution was used for analysis where incidence rate was exponentiated LS mean & incidence rate ratio (IRR) was exponentiated LS mean difference from placebo. Reported p-value is adjusted for multiplicity; IRR = 0.48, 95% CI 2-sided [0.25 to 0.93]
Statistical Analysis 2: Comparison: Placebo vs TAK-861 2 mg BID; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.034, GEE — The GEE model featuring a negative binomial distribution was used for analysis where the incidence rate was the exponentiated LS mean and the IRR was the exponentiated LS mean difference from placebo. Reported p-value is adjusted for multiplicity; IRR = 0.36, 95% CI 2-sided [0.16 to 0.79]
Statistical Analysis 3: Comparison: Placebo vs TAK-861 2 mg and 5 mg; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.003, GEE — [p-value comment as in outcome 3, analysis 2]; IRR = 0.28, 95% CI 2-sided [0.13 to 0.60]
Statistical Analysis 4: Comparison: Placebo vs TAK-861 7 mg QD; [analysis description as in outcome 3, analysis 1]; Test type: Superiority; p = 0.250, GEE — [p-value comment as in outcome 3, analysis 2]; IRR = 0.67, 95% CI 2-sided [0.35 to 1.29]

4. Secondary Outcome: Number of Participants With at Least One Treatment-emergent Adverse Event (TEAE)
Description: An adverse event (AE) was defined as any untoward medical occurrence in a clinical study participant, temporally associated with the use of the study intervention, whether or not the occurrence was considered related to the study intervention. An AE can therefore be any unfavorable and unintended sign (example, a clinically significant abnormal laboratory finding), symptom, or disease temporally associated with the use of a drug, whether or not it is considered related to the drug. A TEAE was defined as an AE with an onset that occurred after receiving study drug.
Time Frame: From first dose of the study drug up to end of the study (up to 3 months)
Population: Safety Analysis Set included all participants who received at least one dose of study drug.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg and 5 mg | TAK-861 7 mg QD
Number analyzed (Participants) | 22 | 23 | 21 | 23 | 23
Participants | 7 | 13 | 15 | 21 | 21

ADVERSE EVENTS:
Time Frame: From first dose of the study drug up to end of the study (up to 3 months)
Description: Safety Analysis Set included all participants who received at least one dose of study drug.
Groups:
- TAK-861 2 mg/5 mg: Participants received TAK-861 2 mg followed by the 5 mg dose, orally, from Days 1 to 56.
Arm/Group | Placebo | TAK-861 0.5 mg BID | TAK-861 2 mg BID | TAK-861 2 mg/5 mg | TAK-861 7 mg QD
All-Cause Mortality (participants affected / at risk) | 0/22 | 0/23 | 0/21 | 0/23 | 0/23
Serious Adverse Events (participants affected / at risk) | 0/22 | 0/23 | 0/21 | 1/23 | 0/23
Other Adverse Events (participants affected / at risk) | 5/22 | 11/23 | 15/21 | 20/23 | 20/23
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | TAK-861 0.5 mg BID (N=23) | TAK-861 2 mg BID (N=21) | TAK-861 2 mg/5 mg (N=23) | TAK-861 7 mg QD (N=23)
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=22) | TAK-861 0.5 mg BID (N=23) | TAK-861 2 mg BID (N=21) | TAK-861 2 mg/5 mg (N=23) | TAK-861 7 mg QD (N=23)
Constipation (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Decreased appetite (Metabolism and nutrition disorders) | 0 | 0 | 0 | 1 | 2
Dizziness (Nervous system disorders) | 0 | 0 | 0 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 2 | 0 | 0
Headache (Nervous system disorders) | 1 | 1 | 3 | 2 | 2
Increased appetite (Metabolism and nutrition disorders) | 1 | 0 | 2 | 1 | 1
Insomnia (Psychiatric disorders) | 1 | 5 | 10 | 13 | 15
Micturition urgency (Renal and urinary disorders) | 1 | 5 | 4 | 12 | 9
Middle insomnia (Psychiatric disorders) | 0 | 1 | 0 | 3 | 0
Nasopharyngitis (Infections and infestations) | 0 | 0 | 2 | 2 | 2
Nausea (Gastrointestinal disorders) | 0 | 0 | 0 | 0 | 2
Pollakiuria (Renal and urinary disorders) | 1 | 3 | 7 | 7 | 12
Pyrexia (General disorders) | 0 | 2 | 0 | 0 | 0
Salivary hypersecretion (Gastrointestinal disorders) | 1 | 2 | 2 | 6 | 2

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2022-08-17): https://cdn.clinicaltrials.gov/large-docs/03/NCT05687903/Prot_000.pdf
  • Statistical Analysis Plan (2023-12-11): https://cdn.clinicaltrials.gov/large-docs/03/NCT05687903/SAP_001.pdf